CLINICAL TRIAL: NCT00824070
Title: An Open-Label, Randomized Assessment of the Concentrations of Besifloxacin, Moxifloxacin, or Gatifloxacin in the Aqueous Humor of Subjects After a Single Topical Dose
Brief Title: Assessment of the Concentrations of Besifloxacin, Moxifloxacin, or Gatifloxacin in the Aqueous Humor of Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 575
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2010-10-29 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Cataract Extraction
Keywords: Bioavailability
MeSH Terms: interventions — besifloxacin; Moxifloxacin; Gatifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Besifloxacin (Experimental): Besifloxacin ophthalmic suspension
  Interventions: Drug: Besifloxacin hydrochloride
- Moxifloxacin (Active Comparator): Vigamox (moxifloxacin ophthalmic solution, 0.5%)
  Interventions: Drug: moxifloxacin hydrochloride
- Gatifloxacin (Active Comparator): Zymar (gatifloxacin ophthalmic solution, 0.3%)
  Interventions: Drug: gatifloxacin

INTERVENTIONS:
Drug: Besifloxacin hydrochloride — Instill besifloxacin study medication in the study eye prior to making an incision for cataract extraction surgery.
  Other Names: Besivance
  Arms: Besifloxacin
Drug: moxifloxacin hydrochloride — Instill moxifloxacin study medication in the study eye prior to making an incision for cataract extraction surgery.
  Other Names: Vigamox
  Arms: Moxifloxacin
Drug: gatifloxacin — Instill gatifloxacin study medication in the study eye prior to making an incision for cataract extraction surgery.
  Other Names: Zymar
  Arms: Gatifloxacin

SUMMARY:
This study is being conducted to assess the concentration of besifloxacin, moxifloxacin, or gatifloxacin in aqueous humor samples collected following topical instillation of the associated formulation in subjects undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are a candidate for a routine, uncomplicated, primary cataract extraction.
* Subjects who, in the Investigator's opinion, have potential for postoperative best corrected Snellen visual acuity of at least 20/200 in the study eye.

Exclusion Criteria:

* Subjects who have a known sensitivity, contraindication, or allergy to the study medication(s) or their components.
* Subjects who had any corneal refractive surgery in the study eye.
* Subjects who have a history or presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the result of the study.
* Subjects who had ocular surgery in the study eye, including laser procedures, within the past 6 months.
* Subjects who have taken any topical ocular medication in the study eye, other than those required by the protocol and permitted for surgery, during the 24 hours prior to the study medication being instilled.
* Subjects who use any antibiotics (e.g., systemic or topical) within the 7 days prior to the surgery date.
* Subjects who are monocular.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donnefeld, Principal Investigator — Ophthalmic Consultants of Long Island
Locations (1):
- Ophthalmic Consultants of Long Island, Rockville Centre, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted a 6 sites in the US. This was a single dose study with first patient enrollment on 2/2/2009 and last patient visit was 7/9/2009.
Pre-assignment Details: 105 subjects were screened at Visit 1 and qualified subjects returned on the day of surgery (Visit 2).
Period: Overall Study
Arm/Group | Besifloxacin | Moxifloxacin | Gatifloxacin
Started | 34 | 35 | 36
Completed | 34 | 35 | 36
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Besifloxacin | Moxifloxacin | Gatifloxacin | Total
Number analyzed (Participants) | 34 | 35 | 36 | 105
Age, Customized [Number; unit: participants]
  <60 years | 4 (8.1) | 4 (9.9) | 5 (9.6) | 13
  60-69 years | 15 | 7 | 10 | 32
  70-79 years | 11 | 19 | 14 | 44
  >/= 80 | 4 | 5 | 7 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 20 | 59
  Male | 16 | 14 | 16 | 46
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 31 | 33 | 34 | 98
  Non-Caucasian | 3 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Aqueous Humor Drug Concentration.
Description: An aqueous humor specimen was collected from the study eye for determination of drug concentration 60 min after study drug instillation.
Time Frame: Visit 2, 1-14 days following screening visit
Population: Statistical Analysis of AH Drug Concentration. Modified intent to treat population (mITT). Subjects with non-missing data.
Measure: Mean (Standard Deviation); unit: µg/mL
Units Other Than Participants: eyes
Arm/Group | Besifloxacin | Moxifloxacin | Gatifloxacin
Number analyzed (Participants) | 32 | 35 | 34
Number analyzed (eyes) | 32 | 35 | 34
µg/mL | 0.1349 (0.5820) | 0.6681 (0.4980) | 0.1251 (0.07624)

ADVERSE EVENTS:
Time Frame: Single ocular administration
Arm/Group | Besifloxacin | Moxifloxacin | Gatifloxacin
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/36

LIMITATIONS AND CAVEATS:
All drug concentrations were significantly below MIC90 values for relevant staphylococcal species.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee and the Investigator(s) are completed. The results of the study may be published or presented by the Investigator(s)after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.